CLINICAL TRIAL: NCT05008250
Title: Efficacy and Safety of Metoprolol Tartrate Tablets Combined With Chinese Traditional Medicine on Premature Ventricular Complex: a Multicenter, Randomized, Double-blind, Parallel Controlled Clinical Study.
Brief Title: Efficacy and Safety of Metoprolol Tartrate Tablets Combined With Chinese Traditional Medicine on Premature Ventricular Complex.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Tianjin Lerentang factory (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013019
Record Dates: First submitted 2021-07-25; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-07

CONDITIONS: Premature Ventricular Contraction
MeSH Terms: conditions — Ventricular Premature Complexes | interventions — Metoprolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Prior to the start of the study, the sponsor (or contract research organization) and statistician will make masking of the research drugs. The statistician in this study used statistical software to generate random coding table according to the method of stratified block randomization. Personnel who have no involvement in this study will paste the corresponding drug number on the drug packaging according to the random coding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Metoprolol tartrate (25 mg twice per day, orally) plus TMYXP (40 pills twice per day, orally). the treatment duration is 8 weeks.
  Interventions: Drug: Tongmai Yangxin Pill (TMYXP); Drug: metoprolol tartrate
- control group (Placebo Comparator): Metoprolol tartrate (25 mg twice per day, orally) plus placebo (40 simulated pills twice per day, orally). The treatment is 8 weeks.
  Interventions: Drug: metoprolol tartrate; Drug: placebo

INTERVENTIONS:
Drug: Tongmai Yangxin Pill (TMYXP) — TMYXP is a Chinese patent medicine developed by many years of clinical practice experience. The ingredients of TMYXP are Radix Rehmanniae, Caulis Spatholobi, Polygonum Multiflorum, Colla Corii Asini, Ophiopogonis, Tortoise Shell (vinegar), Radix Codonopsis, Cassia Twig, Jujube, Schisandra Fruit, and Licorice Root. It has the effect of invigorating Qi, nourishing Yin, dredging the pulse, and relieving pain. It is used in treatment of Qi and Yin deficiency syndromes caused by coronary heart disease, angina pectoris, and arrhythmia.
  Metoprolol tartrate (a heart-selective β-blocker) is a class II antiarrhythmic medication that decreases the ventricular rate of supraventricular tachyarrhythmias by inhibition of atrioventricular conduction.
  Arms: study group
Drug: metoprolol tartrate — metoprolol tartrate (a heart-selective β-blocker) is a class II antiarrhythmic medication that decreases the ventricular rate of supraventricular tachyarrhythmias by inhibition of atrioventricular conduction.
  Other Names: metoprolol; betaloc
Drug: placebo — simulated pills
  Arms: control group

SUMMARY:
Objective: investigators investigated the effects of metoprolol tartrate plus Tongmai Yangxin Pill on premature ventricular complexes and cardiac function in patients with premature ventricular complex.

Methods: In total, 584 participants with premature ventricular complex will be randomly assigned (at a 1:1 ratio) into two groups: study group (metoprolol tartrate [25 mg twice per day, orally] plus Tongmai Yangxin Pill [40 pills twice per day, orally]) and control group (metoprolol tartrate [25 mg twice per day, orally] plus placebo [40 simulated pills twice per day, orally]). The total treatment period is 8 weeks.

Efficacy endpoints and safety assessment:

Primary efficacy endpoints are as follows: change in 24-h number of PVCs after treatment and effective rate of 24-h number of PVCs after treatment. Secondary efficacy endpoints are as follows: change in New York Heart Association classification; total effective rate of comprehensive effect; change in high-sensitivity C-reactive protein level; and change in echocardiography parameters (i.e., left ventricular ejection fraction, left ventricular end diastolic dimension, E/A, cardiac index, cardiac output, and stroke volume).

ELIGIBILITY:
Inclusion Criteria:

* Lown PVC grade, II-IVA;
* in patients with coronary heart disease and comorbid PVC or non-organic heart disease, the PVC frequency was 3000-30000 times/24 h;
* New York Heart Association grade, I or II;
* ejection fraction, ≥45%;
* written informed consent to participate in the trial.

Exclusion Criteria:

* presence of bradyarrhythmia (<50 beats/min), including sinus syndrome and atrioventricular block (second or third degree atrioventricular block);
* presence of persistent ventricular tachycardia, non-persistent ventricular tachycardia, and/or persistent atrial fibrillation;
* presence of severe PVC requiring treatment with other antiarrhythmic drugs; -presence of drug-induced, electrolyte-induced, or acid-base-induced arrhythmia;
* presence of uncontrolled or severe hypertension (e.g., grade ≥3 hypertension);
* presence of uncontrolled diabetes; presence of alanine aminotransferase or aspartate aminotransferase level ≥1.5-fold above the upper limit of normal, urea nitrogen level ≥1.2-fold above the upper limit of normal, and/or blood creatinine above the upper limit of normal;
* presence of severe respiratory dysfunction or asthma;
* presence of primary hematopoietic diseases, other systemic diseases (e.g., hyperthyroidism), poor peripheral circulation perfusion, severe peripheral vascular diseases, and/or PVC with unknown etiology;
* presence of allergic constitution, mental disorder, alcoholism, and/or smoking habit;
* pregnancy or lactation;
* ongoing β-blocker treatment or contraindications to β-blocker treatment; -participation in other clinical trials within the prior 3 months;
* and other reasons for lack of suitability to participate in this study, as determined by the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in 24-h number of PVCs after 8-week treatment | 8 weeks
Effective rate of 24-h number of PVCs after 8-week treatment. | 8 weeks
  the definition of "effective" is, premature ventricular complex decreased by 50%-70% compared with baseline in the Holter result.

SECONDARY OUTCOMES:
change in New York Heart Association (NYHA) classification | 8 weeks
  Marked effective NYHA improvement was defined as reduction of NYHA grade by ≥2; effective NYHA improvement was defined as reduction of NYHA grade by 1; non-effective NYHA improvement was defined as no change or elevation of NYHA grade.
total effective rate of comprehensive effect | 8 weeks
  Total effective rate of comprehensive effect was defined as total symptom score; clinical recovery was defined as significant improvement of clinical symptoms and reduction of symptom score by ≥90%.
change in high-sensitivity C-reactive protein level | 8 weeks
change in echocardiography parameter left ventricular ejection fraction | 8 weeks
change in echocardiography parameter left ventricular end diastolic dimension | 8 weeks
change in echocardiography parameter E/A | 8 weeks
change in echocardiography parameter cardiac index | 8 weeks
change in echocardiography parameter cardiac output | 8 weeks
change in echocardiography parameter stroke volume | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Qi Hua, PhD, Principal Investigator — Xuanwu Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No